CLINICAL TRIAL: NCT04668001
Title: Transcranial Photobiomodulation With Near-Infrared Light for Language in Individuals With Down Syndrome
Acronym: TransPhoM-DS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Paolo Cassano, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020P003611
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Down Syndrome
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Near-Infrared Transcranial Photobiomodulation (tPBM-NIR) (Experimental): tPBM-NIR involves the use of a device that administers near-infrared light over the scalp. The light activates target brain regions.
  Interventions: Device: Near-Infrared Transcranial Photobiomodulation
- Sham Transcranial Photobiomodulation (tPBM-Sham) (Placebo Comparator): tPBM-Sham involves the use of an identical device to tPBM-NIR but does not administer near-infrared light. It mimics the sensation by applying heat but does not actually activate target regions of the brain
  Interventions: Device: Sham Transcranial Photobiomodulation

INTERVENTIONS:
Device: Near-Infrared Transcranial Photobiomodulation — tPBM-NIR involves the use of a device that administers near-infrared light over the scalp. The light activates target brain regions.
  Other Names: tPBM-NIR
  Arms: Near-Infrared Transcranial Photobiomodulation (tPBM-NIR)
Device: Sham Transcranial Photobiomodulation — tPBM-Sham involves the use of an identical device to tPBM-NIR but does not administer near-infrared light. It mimics the sensation by applying heat but does not actually activate target regions of the brain
  Other Names: tPBM-Sham
  Arms: Sham Transcranial Photobiomodulation (tPBM-Sham)

SUMMARY:
The aim of this study is to better understand the effects of transcranial photobiomodulation (tPBM) on neural oscillations of individuals diagnosed with Down syndrome.

DETAILED DESCRIPTION:
This study will compare the effect of tPBM to sham tPBM on gamma neural oscillations in the brain as assessed by EEG, and on language, attention and memory as assessed by neuropsychological testing. Participants will be randomized to either tPBM with near-infrared light (tPBM-NIR) or tPBM-Sham and will undergo 18 treatments (3 treatments per week for 6 weeks) in addition to baseline, short-term and long- term follow up visits.

ELIGIBILITY:
Inclusion criteria for this study include:

1. adult men and women between the ages of 16 and 35
2. diagnosis of DS (i.e., clinical diagnosis of Trisomy 21 or Complete Unbalanced Translocation of Chromosome 21)

Exclusion criteria for this study include:

1. diagnosis of seizure disorder
2. diagnosis of dementia
3. inability to complete study procedures
4. English as a second language
5. speech as the secondary mode of communication
6. speech of less than two-word utterances
7. changes in medications, augmentative devices, and other intervention two weeks prior to baseline testing and throughout study completion at PI's discretion
8. untreated obstructive sleep apnea (OSA)
9. Participation in other clinical research trials that may influence affect primary outcomes or adherence to the proposed study, as assessed by the PI and the Co-Is
10. candidates who have a current diagnosis of cancer and/or are currently undergoing treatment for cancer
11. history of migraine with an aura in the past 6 months
12. current pregnancy

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in EEG | Baseline to Post-Treatment (~6 weeks)
  Gamma Power (40 Hz) of EEG Signal
Change in Wordless Picture Book | Baseline to Post-Treatment (~6 weeks)
  Standardized narrative sampling tasks that measure intelligibility, vocabulary, syntax and grammar of language
Change in Cambridge Neuropsychological Test Automated Battery | Baseline to Post-Treatment (~6 weeks)
  Reaction Time, Paired Associative Learning, and Motor Screening Task subtests

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Cassano, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital at the Charlestown Navy Yard, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No